CLINICAL TRIAL: NCT00715559
Title: An Open-Label Study of Cysteamine Bitartrate in Treatment-Resistant Major Depression
Brief Title: Cysteamine Therapy for Major Depressive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in resources available for study procedures.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO # 07-0478
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2011-06-16 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder, depression; neurotrophic; brain-derived neurotrophic factor; antidepressant; cysteamine
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cysteamine bitartrate (Experimental): Participants received cysteamine bitartrate by mouth up to 300 mg three times daily.
  Interventions: Drug: cysteamine bitartrate

INTERVENTIONS:
Drug: cysteamine bitartrate — All enrolled participants will begin open treatment with cysteamine on the first visit of the experimental period (after screening, medical clearance and medication washout period if necessary). The dosing schedule is a flexible regimen starting at 150 mg PO three times daily. After one week, patients without intolerable side effects will increase the dose to 300 mg three times daily. The titration schedule will continue up to a maximum of 1800 mg a day. In case of adverse events, the investigator may decrease the dose by 150 mg daily.

SUMMARY:
The purpose of this study is to determine whether cysteamine bitartrate, an FDA-approved drug for a non-psychiatric condition, is safe and effective for the treatment of major depression.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a chronic, disabling illness affecting about 17% of the general population. Despite advances in treatment, about two-thirds of patients fail to respond to an initial trial of pharmacotherapy. Brain-derived neurotrophic factor (BDNF) is a neural growth-promoting polypeptide found in the central nervous system, and has been implicated in the pathophysiology and potential treatment of MDD. A multitude of studies have shown low levels of BDNF in subjects with MDD, which have normalized after treatment with an antidepressant. Traditional antidepressants such as serotonin reuptake inhibitors may increase BDNF via an indirect intracellular pathway. The current study drug, cysteamine bitartrate (Cystagon), is FDA approved for the treatment nephropathic cystinosis and has been shown to increase BNDF in neuronal tissue, and to stimulate cell growth. Cysteamine has already been investigated in humans as a potential treatment for Huntington's Disease. Given the evidence of decreased levels in major depression, and subsequent increase post-treatment with antidepressants, BDNF may play a key role in developing novel treatments for patients who have failed conventional agents. Therefore, drugs that can demonstrably increase central BDNF, such as cysteamine, may have significant potential as novel antidepressant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 21-65 years of age.
2. Female subjects who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or must be using a medically accepted means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative serum B-HCG at pre-study.
3. Subjects must fulfill DSM-IV criteria for Major Depression without psychotic features, based on clinical assessment by a study psychiatrist and confirmed by a structured diagnostic interview, the Structured Clinical Interview for DSM-IV TR Axis I Disorders, (SCID-P).
4. Subjects have a history of at least one previous episode of depression prior to the current episode (recurrent major depressive disorder) or have chronic major depressive disorder (at least two years' duration).
5. Subjects have not responded to an adequate trial of one antidepressant in the current episode as determined by Antidepressant Treatment History Form (ATHF) criteria (score > 3) (Sackeim 2001)
6. Subjects must have an initial score of ³ 32 on the IDS-C at both Visit 1 and Visit 2.
7. Each subject must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document.
8. Current major depressive episode is of at least 4 weeks duration

Exclusion Criteria:

1. Presence of psychotic features, diagnosis of schizophrenia or any other psychotic disorder, or bipolar disorder/cyclothymia as defined in the DSM-IV.
2. Lifetime histories of autism, mental retardation, pervasive developmental disorders, OCD, or Tourette's
3. Current Eating Disorder
4. Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for nicotine or caffeine) within the preceding 3 months.
5. Female subjects who are either pregnant or nursing.
6. Serious, unstable illnesses including hepatic, renal, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease.
7. Hypersensitivity to cysteamine or penicillamine
8. Past history of severe gastrointestinal disease (including peptic ulcers or inflammatory bowel disease), or current gastroesophageal reflux disease
9. Subjects with a history of neutropenia or medication-induced blood dyscrasia.
10. Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG.
11. Subjects with uncorrected hypothyroidism or hyperthyroidism.
12. Subjects with one or more seizures without a clear and resolved etiology.
13. Treatment with a reversible MAOI within 2 weeks prior to Visit 2.
14. Treatment with fluoxetine within 4 weeks prior to Visit 2.
15. Treatment with any other concomitant medication not allowed 14 days prior to study Visit 2.
16. Treatment with clozapine or ECT within 3 months prior to study Visit 2.
17. Judged clinically to be at serious suicidal or homicidal risk.
18. Participation in a clinical trial of another investigational drug within 1 month prior to study entry.
19. Patients starting hormonal treatment (e.g., estrogen) in the last 3 months prior to visit 1.
20. Psychotherapy or nonpharmacological antidepressant treatments (e.g. light therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3 participants were recruited between June 2007 and May 2009.
Pre-assignment Details: Participants with major depression were enrolled if they had previously failed to respond to at least one FDA-approved antidepressant. There are no prospective treatment or lead-in and the study was conducted open-label.
Groups:
- Cysteamine Bitartrate: Study participants received cysteamine bitartrate by mouth up to 300 mg three times daily
Period: Overall Study
Arm/Group | Cysteamine Bitartrate
Started | 3
Completed | 2
Not Completed | 1
Not completed — medication not tolerated - nausea | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: This scale measures depression severity. It ranges from a score of 0 to 60, with higher score indicating higher level of depression severity.
Time Frame: 8 weeks
Population: Mean MADRS score at end of treatment (LOCF) in 3 participants treated with cysteamine bitartrate.
Measure: Mean (Standard Deviation); unit: scale score
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 3
scale score | 27 (3)

2. Secondary Outcome: Clinical Global Impression Scales for Severity (CGI-S) and Improvement (CGI-I)
Description: This set of scales measures "global" improvement in a patient's level of symptoms, without reference to a particular condition (ie depression). GCI-S is a measure of severity, which ranges from 0 (not ill) to 7 (severely ill). CGI-I is a measure of change, with a score of 4 indicating no change, 1 indicating very much improved and 7 indicating very much worse.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: scale score
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 3
scale score | 4 (0)

3. Secondary Outcome: Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR16)
Description: This is a self-report which measures the level of depression severity. I ranges from 0 (no illness) to 27 (severe illness).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: scale score
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 3
scale score | 13.3 (2.9)

4. Secondary Outcome: Systematic Assessment for Treatment Emergent Effects (SAFTEE)
Description: The SAFTEE is used to measure somatic and other symptoms which may arise during the course of a clinical trial. This is a non-quantitative instrument that does not yield a numeric score. Instead, it provides study subjects the opportunity to check off symptoms listed on a checklist and indicate if the severity of the symptoms is "mild" "moderate" or "severe." The reported values represent symptoms that were indicated at any point during the 8 week trial at a level of "moderate" or "severe" that also represented a change from a baseline-line pre-intervention SAFTEE assessment.
Time Frame: weekly, for 8 weeks
Population: Study participants were assessed for side effects or adverse events with the SAFTEE at each study visit over the 8 week trial.
Measure: Mean (Standard Deviation); unit: symptoms
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 3
symptoms | 24.3 (17.5)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events are recorded with the SAFTEE at each weekly visit during the 8 week study. All items reported here are endorsed with a severity greater than mild (e.g. moderate or severe) and represent a change from baseline.
Arm/Group | Cysteamine Bitartrate
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cysteamine Bitartrate (N=3)
Numbness or tingling (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Drooling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 1 (1)
loss of sexual interest (Reproductive system and breast disorders) | 1 (1)
appetite decrease (Gastrointestinal disorders) | 1 (1)
word finding difficulty (Nervous system disorders) | 1 (1)
bruising (Vascular disorders) | 1 (1)
hot flashes (Endocrine disorders) | 1 (1)
apathy (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes